CLINICAL TRIAL: NCT06546852
Title: The Effect of Fluid Training Given to Hemodialysis Patients on Interdialytic Fluid Intake and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beykent (Other)
Responsible Party: Principal Investigator, Ülkü YILMAZ, phd internal diseases nurse, University of Beykent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 29 temmuz
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Education; Nursing Caries
Keywords: education
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The study sample, conducted with an experimental design, consisted of 71 patients (36 experimental and 35 control) who received dialysis treatment in a private dialysis centre affiliated with the Istanbul Provincial Health Directorate.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will be informed about the purpose and method of the research and will be informed in writing.
  Informed consent was obtained. Patient Tracking Form, which is a data collection tool, The researcher filled out the Fluid Restriction Scale in Hemodialysis Patients through face-to-face interviews with the patients.
  The results of the biochemical parameters requested by the physician were recorded. Later Patients will be given a 15-20 minute individual session on fluid restriction in chronic renal failure.
  A training and education booklet was provided. At the end of the training, the Fluid Restriction Scale in Hemodialysis Patients was applied to the experimental group as a posttest.
  Interventions: Behavioral: education
- Control group (No Intervention): As for the control group, Information was given about the purpose and method of the research, and a written Informed consent was obtained. Data collection tools: Patient Follow-up Form, Hemodialysis patients fluid restriction scale The researcher completed it during face-to-face interviews with the patients. At the end of the follow-up period, the hemodialysis patients completed the fluid restriction scale as a final test.

INTERVENTIONS:
Behavioral: education — Patient education will be provide
  Other Names: Patient education will be provide
  Arms: Experimental group

SUMMARY:
The research evaluated the effect of nutrition and fluid restriction training on interdialytic fluid intake and intradialytic hypotension in hemodialysis patients. The study sample, conducted with an experimental design, consisted of 71 patients (36 experimental and 35 control) who received dialysis treatment in a private dialysis centre affiliated with the Istanbul Provincial Health Directorate.

DETAILED DESCRIPTION:
The research evaluated the effect of nutrition and fluid restriction training on interdialytic fluid intake and intradialytic hypotension in hemodialysis patients. The study sample, conducted with an experimental design, consisted of 71 patients (36 experimental and 35 control) who received dialysis treatment in a private dialysis centre affiliated with the Istanbul Provincial Health Directorate. Fluid Control Scale in Hemodialysis Patients (HHSÖ), Blood Pressure Control Form, Bioimpedance Analysis, Bioimpedance Analysis Compliance Form, Things to Consider Before Bioimpedance Analysis, and Nutrition Booklet for Dialysis Patients were used to collect the data. Parametric methods were used to analyze the data. Differences between the proportions of categorical variables in independent groups were analyzed with Chi-Square and Fisher's exact tests. The t-test was used to compare quantitative continuous data between two independent groups. A dependent group t-test was used to compare intra-group measurements.

After randomization of the experimental and control groups, both groups were measured with the BCM (Fresenius Medical Care Body Composition Monitor) device. The experimental group was given face-to-face fluid restriction training in line with the Nutrition Booklet for Dialysis Patients. At the end of the second month, BCM was measured again in both groups. During the follow-up of the experimental group, training was repeated according to the needs of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* volunteering
* good communication
* chronic kidney failure
* no amputation
* hemodialysis 3 days a week

Exclusion Criteria:

* Heart battery
* dialysis 2 days a week
* more than 200ml of urine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Complying with fluid restriction | 14 weeks,
  Thanks to the training given, patients consume less fluid. posttests were performed usingthe fluid control scale on Hemdodialysis patients.
  The lowest score from the scale is 24 and the highest score is 72. from scale As the score increases, patients' compliance with fluid control also increases.

CONTACTS AND LOCATIONS:
Overall Officials: ülkü yılmaz, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Ülkü Yılmaz, Istanbul, Turkey (Türkiye)